CLINICAL TRIAL: NCT06140849
Title: Evaluation of Artificial Intelligence Models for Diagnosis of Anterior Open Bite Malocclusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Heba El-Sayed Kamel Akl, Lecturer at Orthodontic Department- Faculty of Dentistry, Cairo University
Other Study IDs: 2107765
Record Dates: First submitted 2023-11-15; First posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-11

CONDITIONS: Artificial Intelligence; Open Bite
MeSH Terms: conditions — Open Bite

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: artificial intelligence model — artificial intelligence model of anterior open bite diagnosis

SUMMARY:
Building artificial intelligence models for diagnosis of anterior open bite malocclusion

DETAILED DESCRIPTION:
The study aims at creating artificial intelligence models, with the input being the pre-treatment photographs and radiographs of open bite patients that are routinely taken for diagnosis and treatment planning. The output of the AI model will be the type and phenotype of anterior open bite. The photographs and radiographs with highest quality will be arranged in certain standardized templates to facilitate the machine learning process.

ELIGIBILITY:
Inclusion Criteria:

* anterior open bite

Exclusion Criteria:

* craniofacial syndromes, previous orthodontic treatment, poor quality records

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any patient with anterior open bite of any type and severity will be included in the study
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
the efficiency of artificial intelligence (AI) model in diagnosis of anterior open bite | 8 months
  The percentage of agreement between the AI model result and the actual diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Yehya Mostafa, DDS., PhD, Study Director — Cairo
Locations (1):
- Orthodontic Department, Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided